CLINICAL TRIAL: NCT03224247
Title: Comparison Between Vertical Splitting Versus Transverse Cutting of Muscle Layer in Lower Segment Cesarean Sections to Avoid Uterine Vessels Injury: a Randomized Controlled Trial
Brief Title: Vertical Splitting of Muscle Layer in Lower Segment Cesarean Sections to Avoid Uterine Vessels Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abass, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Vertical splitting in CS
Record Dates: First submitted 2017-07-15; First posted 2017-07-21 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Cesarean Section Complications
Keywords: vertical splitting; Cesarean Section Complications; uterine vessels; injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transverse splitting (Active Comparator): transverse cutting and/or pulling of lower uterine segment during lower segment cesarean section.
  Interventions: Procedure: Transverse cutting
- Vertical splitting (Active Comparator): vertical splitting,of lower uterine segment during lower segment cesarean section.
  Interventions: Procedure: vertical splitting

INTERVENTIONS:
Procedure: Transverse cutting — Transverse cutting and/or pulling.of lower uterine segment during lower cesarean section extending the uterine incision laterally.
  Arms: Transverse splitting
Procedure: vertical splitting — vertical splitting of lower uterine segment during lower cesarean section making the direction of traction up and downward instead of being laterally and we suppose that this will allow the tissues to split along their natural arrangement, decreasing the probability of extension of the wound into the uterine vessels, thus; decreasing blood loss; operative time and maternal recovery.
  Arms: Vertical splitting

SUMMARY:
Cesarean section is one of the oldest surgical interventions in the history of medicine.Many variations in cesarean section technique have been studied.The investigatory team are aiming to decrease blood loss during cesarean section by vertical splitting versus transverse cutting of muscle layer in lower segment cesarean sections to avoid uterine vessels injury.

DETAILED DESCRIPTION:
Cesarean section is one of the oldest surgical interventions in the history of medicine.Since the first documented cesarean delivery in 1020 AD, various modifications have been made in the technique. It was a surgery performed as a last resort, mostly peri- or post-portem.

Many variations in cesarean section technique have been studied.our study aim is to decrease blood loss during cesarean section through decreasing incidence of uterine vessels injury. The investigator supposed that applying Vertical pull on a small C-shaped incision in the lower uterine segment during cesarean section allows the tissues to split along their natural arrangement, decreasing the probability of extension of the wound into the uterine vessels, thus; decreasing blood loss; operative time and maternal recovery.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section
* No medical disorders during pregnancy ( Hypertension, DM , ..)
* No coagulation disorders either congenital nor acquired.

Exclusion Criteria:

* Urgent or emergency cesarean section.
* Multiple pregnancy.
* Presence of medical disorders during pregnancy ( Hypertension, DM , ..)
* Presence of coagulation disorders either congenital nor acquired.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Uterine vessels injury | 1 minute after extraction of the baby and placenta
  the surgeon performing the cesarean section will detect if injury of uterine vessels occurred or not while extending uterine incision.

SECONDARY OUTCOMES:
uterine incision extension | 2 minutes extraction of the baby and placenta
  the surgeon performing the cesarean section will detect if uterine incision extension occurred or not after extraction of the baby and the placenta.
intra-operative blood loss | before closure of the abdominal wall layer
  blood loss will be assessed by circulating nurse through counting soaked surgical towels and gauze and calculating estimated blood loss in vacation suction system.
postpartum hemorrhage | first 24 hours after delivery
  will be defined by postpartum blood loss of 1000cc
postoperative pain | 2 hours after delivery
  pain scale from 0 to 10 to assess postoperative pain after delivery
postoperative pain | 6 hours after delivery
  pain scale from 0 to 10 to assess postoperative pain at hours 2 after delivery
postoperative pain | 12 hours after delivery
  pain scale from 0 to 10 to assess postoperative pain at hours 2 after delivery
postoperative pain | 24 hours after delivery
  pain scale from 0 to 10 to assess postoperative pain at hours 2 after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Waled Hitler, Prof, Study Director — AinShams University
Locations (1):
- Ahmed Abass, Cairo, Egypt